CLINICAL TRIAL: NCT02256436
Title: A Phase III Randomized Clinical Trial of Pembrolizumab (MK-3475) Versus Paclitaxel, Docetaxel or Vinflunine in Subjects With Recurrent or Progressive Metastatic Urothelial Cancer
Brief Title: A Study of Pembrolizumab (MK-3475) Versus Paclitaxel, Docetaxel, or Vinflunine for Participants With Advanced Urothelial Cancer (MK-3475-045/KEYNOTE-045)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-045; 2014-002009-40 (EudraCT Number); 152903 (Registry Identifier: JAPIC-CTI); MK-3475-045 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-09-29; First posted 2014-10-03 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Urothelial Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Bladder cancer
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Urinary Bladder Neoplasms | interventions — pembrolizumab; Paclitaxel; vinflunine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants receive paclitaxel 175 mg/m^2 intravenously (IV) or docetaxel 75 mg/m^2 IV or vinflunine 320 mg/m^2 IV, on Day 1 of each 3-week cycle (Q3W). Eligible participants who experience disease progression may be able to switch over to receive pembrolizumab 200 mg Q3W for up to 35 treatment administrations (up to approximately 2 years).
  Interventions: Drug: paclitaxel; Drug: vinflunine; Drug: docetaxel
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg IV on Day 1 Q3W. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab 200 mg for up to 17 cycles (up to approximately 1 additional year).
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Drug: paclitaxel — IV infusion
  Arms: Control
Drug: vinflunine — IV infusion
  Arms: Control
Drug: docetaxel — IV infusion
  Arms: Control

SUMMARY:
Participants with metastatic or locally advanced/unresectable urothelial cancer that has recurred or progressed following platinum-based chemotherapy will be randomly assigned to receive Investigator's choice of paclitaxel, docetaxel, or vinflunine (Control), or pembrolizumab. The primary study hypotheses are that pembrolizumab will prolong Overall Survival (OS) and Progression-free Survival (PFS) compared to paclitaxel, docetaxel, or vinflunine.

DETAILED DESCRIPTION:
For the purposes of this study, participants with a programmed cell death-ligand 1 (PD-L1) combined positive score (CPS) ≥10% were considered to have a strongly PD-L1 positive tumor status and participants with PD-L1 CPS ≥1% were considered to have a PD-L1 positive tumor status.

Effective with Amendment 15, eligible participants who are allocated to the Control arm (Investigator's Choice) and experience disease progression will be provided with the opportunity to switch over to receive pembrolizumab 200 mg one time every three weeks (Q3W) for up to two years of treatment.

ELIGIBILITY:
Inclusion criteria:

* Histologically- or cytologically-confirmed diagnosis of urothelial cancer of the renal pelvis, ureter, bladder, or urethra, that is transitional cell or mixed transitional/non-transitional (predominantly transitional) cell type
* Progression or recurrence of urothelial cancer following a first-line platinum-containing regimen (e.g cisplatin, carboplatin) for metastatic or inoperable locally advanced disease; or adjuvant platinum-based therapy following cystectomy for localized muscle-invasive urothelial cancer with recurrence/progression <=12 months following completion of therapy; or neoadjuvant platinum-containing therapy prior to cystectomy for localized muscle-invasive urothelial cancer with recurrence <=12 months following completion of therapy
* No more than 2 prior lines of systemic chemotherapy for metastatic urothelial cancer
* Able to provide tissue for biomarker analysis from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Measureable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate organ function
* Female participants of childbearing potential have a negative urine or serum pregnancy test; or are surgically sterile, or willing to use 2 acceptable methods of birth control, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of pembrolizumab or 180 days after the last dose of paclitaxel, docetaxel, or vinflunine
* Male participants must be willing to use an adequate method of contraception starting with the first dose of study medication through 120 days after the last dose of pembrolizumab or 180 days after the last dose of paclitaxel, docetaxel, or vinflunine

Exclusion criteria:

* Urothelial cancer that is suitable for local therapy administered with curative intent
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to the first dose of trial medication
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or not recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of study Day 1 or not recovered from adverse events due to a previously administered agent
* Prior therapy with all choices of active comparator
* Known additional malignancy that is progressing or requires active treatment with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cancer; or prostate cancer that was identified incidentally following cystoprostatectomy for bladder cancer that is Stage T2N0M0 or lower, Gleason score<= 6, or prostatic-specific antigen (PSA) undetectable
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic or immunosuppressive agents
* Active cardiac disease
* Evidence of interstitial lung disease or active non-infectious pneumonitis
* Active infection requiring systemic therapy
* History of severe hypersensitivity reaction to paclitaxel, docetaxel, or to other drugs formulated with polysorbate 80 or polyoxyethylated castor oil, or to vinflunine or other vinca alkaloids
* Requires ongoing therapy with a medication that is a strong inhibitor or inducer of the cytochrome 3A4 (CYP3A4) enzymes
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of pembrolizumab or 180 days after the last dose of paclitaxel, docetaxel, or vinflunine
* Prior therapy with an anti-programmed cell death 1 (PD-1) or anti-PD-Ligand 1 agent, or with an agent directed to another co-inhibitory T-cell receptor
* Human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Received a live virus vaccine within 30 days of planned start of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Giannatempo P, Machiels JP, Sassa N, Arranz JA, Fujii Y, Su WP, Keam B, Culine S, Shen YC, Langa JM, Sarid D, Aarts M, Calabro F, Rosenbaum E, Moreno BH, Bavle A, Xu JZ, Rha SY. Impact of Histology on Clinical Outcomes of Pembrolizumab Monotherapy in Patients With Advanced or Metastatic Urothelial Carcinoma in the Phase 3 KEYNOTE-045 and KEYNOTE-361 Trials. Clin Genitourin Cancer. 2025 Apr;23(2):102273. doi: 10.1016/j.clgc.2024.102273. Epub 2024 Nov 15. PMID 40037029
- [Derived] Balar AV, Castellano DE, Grivas P, Vaughn DJ, Powles T, Vuky J, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Necchi A, Petrylak DP, Plimack ER, Xu JZ, Imai K, Moreno BH, Bellmunt J, de Wit R, O'Donnell PH. Efficacy and safety of pembrolizumab in metastatic urothelial carcinoma: results from KEYNOTE-045 and KEYNOTE-052 after up to 5 years of follow-up. Ann Oncol. 2023 Mar;34(3):289-299. doi: 10.1016/j.annonc.2022.11.012. Epub 2022 Dec 6. PMID 36494006
- [Derived] Bellmunt J, de Wit R, Fradet Y, Climent MA, Petrylak DP, Lee JL, Fong L, Necchi A, Sternberg CN, O'Donnell PH, Powles T, Plimack ER, Bajorin DF, Balar AV, Castellano D, Choueiri TK, Culine S, Gerritsen W, Gurney H, Quinn DI, Vuky J, Vogelzang NJ, Cristescu R, Lunceford J, Saadatpour A, Loboda A, Ma J, Rajasagi M, Godwin JL, Homet Moreno B, Grivas P. Putative Biomarkers of Clinical Benefit With Pembrolizumab in Advanced Urothelial Cancer: Results from the KEYNOTE-045 and KEYNOTE-052 Landmark Trials. Clin Cancer Res. 2022 May 13;28(10):2050-2060. doi: 10.1158/1078-0432.CCR-21-3089. PMID 35247908
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Fradet Y, Bellmunt J, Vaughn DJ, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Nam K, Frenkl TL, Perini RF, de Wit R, Bajorin DF. Randomized phase III KEYNOTE-045 trial of pembrolizumab versus paclitaxel, docetaxel, or vinflunine in recurrent advanced urothelial cancer: results of >2 years of follow-up. Ann Oncol. 2019 Jun 1;30(6):970-976. doi: 10.1093/annonc/mdz127. PMID 31050707
- [Derived] Vaughn DJ, Bellmunt J, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Li H, Perini RF, Bajorin DF, de Wit R. Health-Related Quality-of-Life Analysis From KEYNOTE-045: A Phase III Study of Pembrolizumab Versus Chemotherapy for Previously Treated Advanced Urothelial Cancer. J Clin Oncol. 2018 Jun 1;36(16):1579-1587. doi: 10.1200/JCO.2017.76.9562. Epub 2018 Mar 28. PMID 29590008
- [Derived] Rassy EE, Bakouny Z, Aoun F, Haddad FG, Sleilaty G, Assi T, Kattan J. A network meta-analysis of the PD(L)-1 inhibitors in the salvage treatment of urothelial bladder cancer. Immunotherapy. 2018 Jun;10(8):657-663. doi: 10.2217/imt-2017-0190. Epub 2018 Mar 22. PMID 29562804
- [Derived] Bellmunt J, de Wit R, Vaughn DJ, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Poehlein CH, Perini RF, Bajorin DF; KEYNOTE-045 Investigators. Pembrolizumab as Second-Line Therapy for Advanced Urothelial Carcinoma. N Engl J Med. 2017 Mar 16;376(11):1015-1026. doi: 10.1056/NEJMoa1613683. Epub 2017 Feb 17. PMID 28212060
- [Derived] Kim YS, Lee SI, Park SH, Park S, Hwang IG, Lee SC, Sun JM, Lee J, Lim HY. A Phase II Study of Weekly Docetaxel as Second-Line Chemotherapy in Patients With Metastatic Urothelial Carcinoma. Clin Genitourin Cancer. 2016 Feb;14(1):76-81. doi: 10.1016/j.clgc.2015.09.008. Epub 2015 Sep 25. PMID 26454620
- See also: Merck Oncology Clinical trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, 13 participants randomized to receive Control were switched over to receive Pembrolizumab. Per protocol, response/progression or adverse events that occurred during a non-randomized switch-over or second course of pembrolizumab were not counted towards efficacy or safety outcome measures, respectively. These results are for randomized treatment only.
Groups:
- Control: Participants received paclitaxel 175 mg/m^2 intravenously (IV) or docetaxel 75 mg/m^2 IV or vinflunine 320 mg/m^2 IV, on Day 1 of each 3-week cycle (Q3W). Eligible participants who experienced disease progression may have been able to switch over to receive pembrolizumab 200 mg IV Q3W for up to 35 treatment administrations (up to approximately 2 years).
- Pembrolizumab: Participants received pembrolizumab 200 mg IV on Day 1 Q3W. Eligible participants who stopped pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab 200 mg IV Q3W for up to 17 cycles (up to approximately 1 additional year).
Period: Overall Study
Arm/Group | Control | Pembrolizumab
Started | 272 | 270
Treated | 255 | 266
Switched Over to Pembrolizumab | 13 | 0
Completed | 0 | 0
Not Completed | 272 | 270
Not completed — Adverse Event | 9 | 14
Not completed — Death | 216 | 208
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 26 | 10
Not completed — Transferred to Extension Study | 11 | 23
Not completed — Did Not Continue on Extension Study | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Pembrolizumab | Total
Number analyzed (Participants) | 272 | 270 | 542
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (9.2) | 66.0 (10.2) | 65.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 202 | 200 | 402

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - All Participants
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 was assessed by blinded independent central review (BICR) in all participants up through the primary analysis database cut-off date of 07-Sep-2016.
Time Frame: Through primary analysis database cut-off date of 07-Sep-2016 (Up to approximately 20 months)
Population: The analysis population consisted of all randomized participants, regardless of whether or not they received study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 272 | 270
Months | 3.3 [2.3 to 3.5] | 2.1 [2.0 to 2.2]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; PFS - All Participants; Test type: Superiority or Other; p = 0.41648, Regression, Cox — One-sided p-value based on stratified log-rank test; Treatment as a covariate stratified by ECOG PS, presence/absence of liver metastases, hemoglobin and time from completion of most recent chemotherapy; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.81 to 1.19]

2. Primary Outcome: Overall Survival (OS) - All Participants
Description: OS was defined as the time from randomization to death due to any cause. The OS was assessed in all participants up through the primary analysis database cut-off date of 07-Sep-2016.
Time Frame: Through primary analysis database cut-off date of 07-Sep-2016 (Up to approximately 20 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 272 | 270
Months | 7.4 (5.1) [6.1 to 8.3] | 10.3 (37.8) [8.0 to 11.8]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; OS - All Participants (Note: ECOG PS=Eastern Cooperative Oncology Group Performance Status); Test type: Superiority or Other; p = 0.00224, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.91]

3. Primary Outcome: PFS Per RECIST 1.1 - Participants With Programmed Cell Death-Ligand (PD-L1) Positive Tumors
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. PFS per RECIST 1.1 was assessed by BICR in all participants who had PD-L1 positive tumors (combined positive score [CPS] ≥1%) up through the primary analysis database cut-off date of 07-Sep-2016.
Time Frame: Through primary analysis database cut-off date of 07-Sep-2016 (Up to approximately 20 months)
Population: The analysis population consisted of all randomized PD-L1 positive participants, regardless of whether or not they received study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 120 | 110
Months | 3.2 [2.2 to 3.4] | 2.1 [2.0 to 2.4]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; PFS - PD-L1 positive participants; Test type: Superiority or Other; p = 0.26443, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.68 to 1.24]

4. Primary Outcome: OS - Participants With PD-L1 Positive Tumors
Description: OS was defined as the time from randomization to death due to any cause. For the purposes of this study, participants with PD-L1 CPS ≥1% were considered to have a PD-L1 positive tumor status. OS was assessed in all participants who had PD-L1 positive tumors (CPS ≥1%) up through the primary analysis database cut-off date of 07-Sep-2016.
Time Frame: Through primary analysis database cut-off date of 07-Sep-2016 (Up to approximately 20 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 120 | 110
Months | 6.9 [4.7 to 8.8] | 11.3 [7.7 to 16.0]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; OS - PD-L1 positive participants; Test type: Superiority or Other; p = 0.00239, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.43 to 0.86]

5. Primary Outcome: PFS Per RECIST 1.1 - Participants With Strongly PD-L1 Positive Tumors
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. PFS per RECIST 1.1 was assessed by BICR in all participants who had strongly PD-L1 positive tumors (CPS ≥10%) up through the primary analysis database cut-off date of 07-Sep-2016.
Time Frame: Through primary analysis database cut-off date of 07-Sep-2016 (Up to approximately 20 months)
Population: The analysis population consisted of all randomized strongly PD-L1 positive participants, regardless of whether or not they received study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 90 | 74
Months | 3.1 [2.2 to 3.4] | 2.1 [1.9 to 2.1]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; PFS - Strongly PD-L1 positive participants; Test type: Superiority or Other; p = 0.23958, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.61 to 1.28]

6. Primary Outcome: OS - Participants With Strongly PD-L1 Positive Tumors
Description: OS was defined as the time from randomization to death due to any cause. For the purposes of this study, participants with a PD-L1 CPS ≥10% were considered to have a strongly PD-L1 positive tumor status. The OS was assessed in all participants who had strongly PD-L1 positive tumors (CPS ≥10%) up through the primary analysis database cut-off date of 07-Sep-2016.
Time Frame: Through primary analysis database cut-off date of 07-Sep-2016 (Up to approximately 20 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 90 | 74
Months | 5.2 [4.0 to 7.4] | 8.0 [5.0 to 12.3]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; OS - Strongly PD-L1 positive participants; Test type: Superiority or Other; p = 0.00483, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.37 to 0.88]

7. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. Participants were monitored for the occurrence nonserious AEs for up to 30 days after last dose of study treatment and for serious AEs for up to 90 days after last dose of study treatment. The number of participants who experienced an AE was reported for each arm.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Number; unit: Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 255 | 266
Participants | 250 | 250

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. Participants were monitored for the occurrence nonserious AEs for up to 30 days after last dose of study treatment and for serious AEs for up to 90 days after last dose of study treatment. The number of participants who discontinued study treatment due to an AE was reported for each arm.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 255 | 266
Participants | 36 | 28

9. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 - Participants With Strongly PD-L1 Positive Tumors
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR was assessed by BICR in participants with strongly PD-L1 positive tumors (CPS ≥10%) up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 90 | 74
Percentage of Participants | 6.7 [2.5 to 13.9] | 20.3 [11.8 to 31.2]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; ORR per RECIST 1.1 - Strongly PD-L1 Positive Participants; Test type: Superiority or Other; p = 0.00061, Miettinen & Nurminen method — One-sided p-value for testing H0: difference in %=0; H1: difference in %>0; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 17.2, 95% CI 2-sided [6.8 to 29.4]

10. Secondary Outcome: ORR Per RECIST 1.1 - Participants With PD-L1 Positive Tumors
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR was assessed by BICR in participants with PD-L1 positive tumors (CPS ≥1%) up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 120 | 110
Percentage of Participants | 8.3 [4.1 to 14.8] | 22.7 [15.3 to 31.7]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; ORR per RECIST 1.1 - PD-L1 Positive Participants; Test type: Superiority or Other; p = 0.00049, Miettinen & Nurminen method — One-sided p-value for testing H0: difference in %=0; H1: difference in %>0; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 15.6, 95% CI 2-sided [6.5 to 25.7]

11. Secondary Outcome: ORR Per RECIST 1.1 - All Participants
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR was assessed by BICR in all participants up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 272 | 270
Percentage of Participants | 11.0 [7.6 to 15.4] | 21.1 [16.4 to 26.5]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; ORR per RECIST 1.1 - All Participants; Test type: Superiority or Other; p = 0.00068, Miettinen & Nurminen method — One-sided p-value for testing H0: difference in %=0; H1: difference in %>0; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 10.0, 95% CI 2-sided [3.9 to 16.2]

12. Secondary Outcome: PFS Per Modified RECIST (mRECIST) - Participants With Strongly PD-L1 Positive Tumors
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per mRECIST, PD was defined was defined as at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. Per mRECIST, confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required for participants remaining on treatment following PD per RECIST 1.1. PFS per mRECIST was assessed by BICR in participants with strongly PD-L1 positive tumors (CPS ≥10%) up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 90 | 74
Months | 3.3 [2.4 to 3.7] | 2.1 [2.0 to 3.7]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; PFS per mRECIST - Strongly PD-L1 Positive Participants; Test type: Superiority or Other; p = 0.07066, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.53 to 1.11]

13. Secondary Outcome: PFS Per mRECIST - Participants With PD-L1 Positive Tumors
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per mRECIST, PD was defined was defined as at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. Per mRECIST, confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required for participants remaining on treatment following PD per RECIST 1.1. PFS per mRECIST was assessed by BICR in participants with PD-L1 positive tumors (CPS ≥1%) up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 120 | 110
Months | 3.3 [2.6 to 3.6] | 2.1 [2.0 to 3.7]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; PFS per mRECIST - PD-L1 Positive Participants; Test type: Superiority or Other; p = 0.08745, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.60 to 1.10]

14. Secondary Outcome: PFS Per mRECIST - All Participants
Description: PFS was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. Per mRECIST, PD was defined as at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. Per mRECIST, confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented was required for participants remaining on treatment following PD per RECIST 1.1. PFS per mRECIST was assessed by BICR in all randomized participants up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 272 | 270
Months | 3.4 [3.1 to 3.8] | 2.2 [2.1 to 3.3]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; PFS per mRECIST - All Participants; Test type: Superiority or Other; p = 0.05328, Regression, Cox — One-sided p-value based on stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.71 to 1.04]

15. Secondary Outcome: ORR Per mRECIST - Participants With Strongly PD-L1 Positive Tumors
Description: ORR per mRECIST was defined as the percentage of participants in the analysis population who had a CR (complete disappearance of all lesions (and no new lesions), with confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented) or a PR (decrease in tumor burden ≥50% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation). ORR per mRECIST was assessed by BICR in participants with strongly PD-L1 positive tumors (CPS ≥10%) up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 90 | 74
Percentage of Participants | 7.8 [3.2 to 15.4] | 24.3 [15.1 to 35.7]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; ORR per mRECIST - Strongly PD-L1 Positive Participants; Test type: Superiority or Other; p = 0.00009, Miettinen & Nurminen method — One-sided p-value for testing H0: difference in %=0; H1: difference in %>0; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 21.5, 95% CI 2-sided [10.1 to 34.2]

16. Secondary Outcome: ORR Per mRECIST - Participants With PD-L1 Positive Tumors
Description: ORR per mRECIST was defined as the percentage of participants in the analysis population who had a CR (complete disappearance of all lesions (and no new lesions), with confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented) or a PR (decrease in tumor burden ≥50% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation). ORR per mRECIST was assessed by BICR in participants with PD-L1 positive tumors (CPS ≥1%) up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 120 | 110
Percentage of Participants | 9.2 [4.7 to 15.8] | 28.2 [20.0 to 37.6]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; ORR per mRECIST - PD-L1 Positive Participants; Test type: Superiority or Other; p = 0.00002, Miettinen & Nurminen method — One-sided p-value for testing H0: difference in %=0; H1: difference in %>0; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 21.0, 95% CI 2-sided [11.1 to 31.5]

17. Secondary Outcome: ORR Per mRECIST - All Participants
Description: ORR per mRECIST was defined as the percentage of participants in the analysis population who had a CR (complete disappearance of all lesions (and no new lesions), with confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented) or a PR (decrease in tumor burden ≥50% relative to baseline confirmed by a consecutive assessment at least 4 weeks after first documentation). ORR per mRECIST was assessed by BICR in all participants up through the final analysis database cut-off date of 26-Oct-2017.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 272 | 270
Percentage of Participants | 11.4 [7.9 to 15.8] | 25.2 [20.1 to 30.8]
Statistical Analysis 1: Comparison: Control vs Pembrolizumab; ORR per mRECIST - All Participants; Test type: Superiority or Other; p = 0.00001, Miettinen & Nurminen method — One-sided p-value for testing H0: difference in %=0; H1: difference in %>0; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 13.8, 95% CI 2-sided [7.4 to 20.3]

18. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 - Participants With Strongly PD-L1 Positive Tumors
Description: For participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. Per protocol, the DOR was to be censored at the date of the last tumor assessment for participants who had progressed or died after 2 or more missed visits, who had started a new anti-cancer treatment, who were lost to follow-up, or who had an ongoing response. DOR was assessed in all participants who had strongly PD-L1 positive tumors (CPS ≥10%) based on BICR and was analyzed using the Kaplan-Meier method.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: The analysis population consisted of all randomized strongly PD-L1 positive participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1, regardless of whether or not they received study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 6 | 15
Months | 4.4 [2.8 to NA] — NA= DOR upper 95% confidence limit was undefined because the DOR rate was not low enough at the time of the cut-off date. | NA [8.2 to NA] — NA= Median DOR was not reached because there were not enough events, DOR upper 95% confidence limit was undefined because the DOR rate was not low enough at the time of the cut-off date.

19. Secondary Outcome: DOR Per RECIST 1.1 - Participants With PD-L1 Positive Tumors
Description: For participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. Per protocol, the DOR was to be censored at the date of the last tumor assessment for participants who had progressed or died after 2 or more missed visits, who had started a new anti-cancer treatment, who were lost to follow-up, or who had an ongoing response. DOR was assessed in all participants who had PD-L1 positive tumors (CPS ≥1%) based on BICR and was analyzed using the Kaplan-Meier method.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: The analysis population consisted of all randomized PD-L1 positive participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1, regardless of whether or not they received study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 10 | 25
Months | NA [2.8 to NA] — NA= Median DOR was not reached because there were not enough events, DOR upper 95% confidence limit was undefined because the DOR rate was not low enough at the time of the cut-off date. | NA [21.8 to NA] — NA= Median DOR was not reached because there were not enough events, DOR upper 95% confidence limit was undefined because the DOR rate was not low enough at the time of the cut-off date.

20. Secondary Outcome: DOR Per RECIST 1.1 - All Participants
Description: For participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. Per protocol, the DOR was to be censored at the date of the last tumor assessment for participants who had progressed or died after 2 or more missed visits, who had started a new anti-cancer treatment, who were lost to follow-up, or who had an ongoing response. DOR was assessed in all participants based on BICR and was analyzed using the Kaplan-Meier method.
Time Frame: Through final analysis database cut-off date of 26-Oct-2017 (Up to approximately 34 months)
Population: The analysis population consisted of all randomized participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1, regardless of whether or not they received study treatment. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Control | Pembrolizumab
Number analyzed (Participants) | 30 | 57
Months | 4.4 [4.0 to 20.3] | NA [15.9 to NA] — NA = Median DOR was not reached because there were not enough events, DOR upper 95% confidence limit was undefined because the DOR rate was not low enough at the time of the cut-off date.

ADVERSE EVENTS:
Time Frame: Through end of trial analysis database cut-off date of 01-Oct-2020 (Up to approximately 71 months)
Description: All-Cause Mortality table includes all randomized participants. Serious and Other AEs include all treated participants according to treatment received. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug excluded as AEs. Thirteen participants randomized to receive Control were switched over to pembrolizumab per protocol and were monitored for AEs separately.
Groups:
- Control Switched Over to Pembrolizumab: Per protocol, participants originally randomized to the Control arm that experienced disease progression were switched over to receive pembrolizumab 200 mg IV on Day 1 Q3W.
Arm/Group | Control | Pembrolizumab | Control Switched Over to Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 230/272 | 224/270 | 9/13
Serious Adverse Events (participants affected / at risk) | 104/255 | 107/266 | 8/13
Other Adverse Events (participants affected / at risk) | 237/255 | 236/266 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=255) | Pembrolizumab (N=266) | Control Switched Over to Pembrolizumab (N=13)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 6 (7) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (16) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 8 (8) | 0 (0) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 3 (3) | 0 (0)
Hyperthermia malignant (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 5 (5) | 2 (2)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (9) | 11 (11) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (13) | 12 (16) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 3 (3) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 5 (5) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (5) | 6 (6) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasoconstriction (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=255) | Pembrolizumab (N=266) | Control Switched Over to Pembrolizumab (N=13)
Anaemia (Blood and lymphatic system disorders) | 86 (139) | 45 (61) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 41 (74) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 11 (11) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 21 (24) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 33 (40) | 32 (37) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16) | 9 (11) | 0 (0)
Constipation (Gastrointestinal disorders) | 79 (105) | 54 (63) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 47 (69) | 43 (72) | 1 (2)
Nausea (Gastrointestinal disorders) | 73 (100) | 56 (62) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 23 (35) | 7 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 34 (47) | 38 (47) | 0 (0)
Asthenia (General disorders) | 52 (67) | 33 (36) | 0 (0)
Fatigue (General disorders) | 85 (107) | 66 (83) | 3 (3)
Influenza like illness (General disorders) | 7 (8) | 10 (14) | 1 (2)
Mucosal inflammation (General disorders) | 18 (24) | 6 (8) | 0 (0)
Oedema peripheral (General disorders) | 39 (48) | 31 (36) | 0 (0)
Pyrexia (General disorders) | 30 (38) | 36 (44) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 15 (23) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 10 (12) | 1 (1)
Urinary tract infection (Infections and infestations) | 27 (30) | 33 (45) | 2 (2)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5) | 14 (15) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 14 (15) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 9 (9) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 4 (4) | 1 (1)
Blood creatinine increased (Investigations) | 13 (16) | 13 (22) | 2 (2)
Neutrophil count decreased (Investigations) | 40 (73) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 8 (11) | 4 (4) | 1 (1)
Weight decreased (Investigations) | 22 (23) | 25 (30) | 1 (1)
White blood cell count decreased (Investigations) | 22 (41) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 53 (65) | 57 (64) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (9) | 9 (10) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (21) | 16 (20) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (16) | 5 (11) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (57) | 30 (35) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 40 (47) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 15 (16) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (24) | 17 (20) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (31) | 24 (28) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 19 (26) | 19 (22) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (16) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 14 (18) | 14 (19) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 31 (43) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 6 (9) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 28 (34) | 2 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 5 (6) | 1 (1)
Delirium (Psychiatric disorders) | 4 (5) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 20 (20) | 19 (22) | 2 (2)
Haematuria (Renal and urinary disorders) | 17 (21) | 30 (43) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 39 (51) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 31 (38) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (5) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (12) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 100 (106) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 17 (19) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (17) | 66 (88) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 18 (19) | 32 (40) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 7 (8) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 14 (19) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT02256436/Prot_SAP_000.pdf